CLINICAL TRIAL: NCT03090204
Title: Strain Analysis as a Right Ventricle Contractility Marker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16-0370
Record Dates: First submitted 2017-03-10; First posted 2017-03-24 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Systolic Function
Keywords: strain; myocarditic deformation imaging; right ventricle (RV); systolic RV function; preload dependence; contractility; intermittent hemodialysis (HDI)
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound measurements (Other): ultrasound measurements of myocardial deformation of free wall right ventricle during a sharp decline of right ventricle preload induced during a session of Intermittent hemodialysis.
  Interventions: Procedure: ultrasound measurements

INTERVENTIONS:
Procedure: ultrasound measurements — ultrasound measurements of myocardial deformation of free wall right ventricle at 4 time points during a session of intermittent hemodialysis : before the intermittent hemodialysis connection, just after starting hemodialysis, after 1 hour of hemodialysis and 5 minutes before restitution

SUMMARY:
The analysis of the systolic function (contractility) of the right ventricle (RV) is fundamental and central in many pathologies in intensive care unit. It can guide physicians in choosing therapeutics. The conventional ultrasound markers of RV function evaluation currently used are influenced by RV loading conditions, impairing their capacity to approximate a true contractility analysis. Myocardial strain imaging is a recent echographic technique that allows, among other things, to evaluate RV systolic function. It is a reproducible index with early variations which, if it proved to be independent pre-load, would help to better appreciate the RV contractility.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* Patients with renal failure treated with intermittent hemodialysis
* Patients who received an information and did not opposed to participate in the study, or, if unconscious patient at the time of inclusion: a person of trust as defined in Article L. 1111-6 of the Public Health Code, failing that, the family or, failing that, a person maintaining stable link, having received information and not opposed to participate in the study.

Exclusion Criteria:

* Patients with heart disease (valvular, ischemic, rhythmic)
* Patients with ejection fraction of left ventricular altered <45%
* Chronic dialysis patients
* Patients referred in Articles L. 1121-5, L.1121-6, L.1121-7, L.1121-8 of the Public Health Code:

  * Pregnant women, parturients or nursing mothers
  * Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care, persons admitted to a health or social institution for purposes other than research
  * Minor Patients
  * Major persons who are subject to a legal protection measure or are unable to express their consent
* Patients not willing to participate in the study
* Patients not affiliated to a social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the change in the Longitudinal strain of the free wall right ventricle | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound

SECONDARY OUTCOMES:
Evaluation of the change in S' right ventricle wave | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound
Evaluation of the change in tricuspid annular plane systolic excursion (TAPSE) | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound
Evaluation of the change in visual left ventricular ejection fraction (LVEF) | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound
Evaluation of the change in mitral E wave | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound
Evaluation of the change in mitral A wave | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound
Evaluation of the change in wave E ' at the lateral mitral ring | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound
Evaluation of the change in systolic fraction of pulmonary venous flow | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  measurements will be performed using an ultrasound device usually used in our center for the hemodynamic monitoring of patients in intensive care by transthoracic cardiac ultrasound
inter individual variability of Longitudinal strain of the free wall right ventricle | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  Each measurement will be performed by two blind operators
intra individual variability of Longitudinal strain of the free wall right ventricle | at baseline, 1 minute after starting hemodialysis, 1 hour after, and 5 minutes before restitution
  Each measurement will be performed by two blind operators

CONTACTS AND LOCATIONS:
Overall Officials: Zoé Schmitt, Principal Investigator — Hôpital de la Croix-Rousse
Locations (2):
- France (2):
  - Hôpital de la Croix Rousse, Lyon
  - Hopital Saint Joseph Saint Luc, Lyon